CLINICAL TRIAL: NCT06996951
Title: Sinonasal Therapies and Histologic Correlations for Patients With Cystic Fibrosis in the Era of Highly Effective Modulator Therapy
Brief Title: Sinonasal Therapies and Histologic Correlations of Patients With Cystic Fibrosis in the Era of Highly Effective Modulator Therapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: American Rhinologic Society (Other)
Responsible Party: Principal Investigator, Elisa Illing, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26204
Record Dates: First submitted 2025-05-14; First posted 2025-05-30 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis (CF); Chronic Rhinosinusitis (CRS)
MeSH Terms: conditions — Cystic Fibrosis | interventions — Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTINUE TOPICAL STEROID NASAL IRRIGATION (Active Comparator): PARTICIPANTS WILL CONTINUE THEIR NASAL TREATMENT WHICH WAS ALREADY PRESCRIBED BY THEIR PHYSICIAN
  Interventions: Drug: CONTINUE NASAL SALINE IRRIGATION WITH OR WITHOUT STEROID
- STOP TOPICAL NASAL TREATMENT (Experimental): PARTICIPANTS IN THIS ARM WILL BE ASKED TO STOP THEIR NASAL TREATMENT
  Interventions: Other: STOP NASAL SALINE IRRIGATION WITH OR WITHOUT STEROID

INTERVENTIONS:
Other: STOP NASAL SALINE IRRIGATION WITH OR WITHOUT STEROID — PATIENT WILL STOP USING NASAL SALINE IRRIGATION WITH OR WITHOUT STEROID
  Arms: STOP TOPICAL NASAL TREATMENT
Drug: CONTINUE NASAL SALINE IRRIGATION WITH OR WITHOUT STEROID — PATIENT WILL CONTINUE USING NASAL SALINE IRRIGATION WITH OR WITHOUT STEROID
  Arms: CONTINUE TOPICAL STEROID NASAL IRRIGATION

SUMMARY:
The investigators are doing this study to discover if it is appropriate for people with Cystic Fibrosis (CF) on highly effective modulator therapy (HEMT) to stop using certain standard Sino nasal therapies such as high-volume nasal saline irrigations, topical nasal steroids, and topical nasal antibiotics. They are also going to study the fluid inside the nose to see if there are changes when stopping these therapies. Right now, they are not sure if it is suggested to stop these treatments when patients begin highly effective modulator therapy (HEMT)

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a widely known genetic disorder causing patients significant sinopulmonary disease. (1) The advent of highly effective modulator therapy (HEMT) has led to tremendous improvements in manifestations of disease in the lungs, sinuses, along with other organ systems, raising the question of whether and how to de-escalate other treatments for the airways. Specifically for CF, no protocols exist for the de-escalation of the most common sinonasal therapies: high-volume nasal saline irrigations, topical nasal steroids, and topical nasal antibiotics. Establishing such protocols would benefit patients by removing these cumbersome medication regimens, reducing the cost of medications, and lowering risks of side effects and complications from therapies that may no longer provide clinical benefit. This study aims to sample the sinonasal environment for inflammatory markers in patients with cystic fibrosis (PwCF )on HEMT and correlate to subjective and objective clinical findings during de-escalation trials from saline nasal irrigations, topical nasal steroids and/or antibiotics.

The investigators will prospectively follow adult cystic fibrosis patients with chronic rhinosinusitis with or without history of sinus surgery currently using CFTR modulator therapy via diagnostic methods (nasal endoscopy, FEV1, BMI) which are standard of care evaluations currently performed at both Rhinologic and Pulmonary visits. Questions regarding health care utilization (antibiotics, steroids, hospital admissions, doctor visits) will be reviewed, which are also part of the standard history taken at patient intake for these visits. Patient reported outcome measures (PROMS) (SNOT-22, Cystic Fibrosis Questionnaire- Revised (CFQ-R), Patient Health Questionnaire-9 (PHQ-9)) are also routinely collected at these Rhinologic and Pulmonary visits, thus patients are accustomed to these items in routine standard of care followups. Upon enrollment to the study after informed consent obtained, the patients will be randomly assigned to continue or stop topical medicated nasal irrigations. Participants will continue the 1-2 times per day they currently perform the saline topical nasal irrigations, or told to discontinue completely.

To better understand the inflammatory microenvironment on and off HEMT therapy, nasal leukosorb analyses will be studied from at 4-week intervals in the PwCF enrolled in aim 1 for the 12-week study period, to determine trends of inflammation for patients in each arm of the de-escalation study. Following protocols established by Rebuli et al, patients will moisten their nostrils with ~100uL of 0.9% sterile normal saline solution, followed by applying a cut sheet of Leukosorb medium of 4x40mm in length into each nostril onto the anterior part of the inferior turbinate. (19) The nostrils will then be clamped with a padded nose clip. The strips will be removed at 2 minutes, and placed into 1.5mL collection tubes and stored at -20 deg C until fluid elution and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Cystic Fibrosis diagnosis on HEMT
* History of chronic rhinosinusitis
* Using topical nasal irrigations +/- additives (steroids, antibiotics)

Exclusion Criteria:

* Below age of 18 years old
* Cystic Fibrosis patient NOT on highly effective modulator therapy
* Pregnant patients
* Not currently using topical nasal irrigations +/- additives (steroids, antibiotics)
* History of sinonasal or nasopharyngeal tumors
* Active sinonasal infection or pulmonary infection
* Admission to hospital for pulmonary exacerbation within last 3 months
* Oral antibiotics within last one month for upper respiratory or lower respiratory infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Lund Kennedy Score | Baseline, 12 weeks
  Nasal Endoscopy will be performed in the clinic to evaluate the sinonasal cavities using the Lund Kennedy scoring system. The Lund-Kennedy endoscopic score grades the severity of chronic rhinosinusitis (CRS) based on findings from five areas: polyps, discharge, edema, scarring, and crusting, with each graded on a scale of 0 to 2 for each nostril, resulting in a total possible score of 20. A higher score indicates more severe disease.
Change in Pulmonary Function Testing | Baseline, 12 weeks
  PULMONARY FUNCTION TESTING WILL BE PERFORMED WITH THE FEV1/FVC , CALCULATED. A lower score means poorer lung function.
Change in Body Mass Index (BMI) | Baseline, 12 weeks
  BMI will be calculated as weight (kg) / height (m)2
Change in Health Care Utilization | Baseline, 12 weeks
  Health Care Utilization will be measured though a grouped analysis for additional doctor visits, hospital admissions, and use of antibiotics and oral steroids.
Change in Sinonasal Outcome Test 22 Questionnaire (SNOT-22) Score | Baseline, 12 weeks
  The SNOT-22 measures nasal symptoms and social/emotional consequences of rhinosinusitis, rated on a scale of 0 (no problem) to 5 (problem is as bad as it can be). Scores may range from 0 to 110, with higher scores indicating worse sinus symptoms
Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Score | Baseline, 12 weeks
  The Cystic Fibrosis Questionnaire-Revised (CFQ-R) is a disease-specific health-related quality of life (HRQOL) measure for children, adolescents and adults with cystic fibrosis (CF). It is a profile measure of HRQOL with several different domains. The Cystic Fibrosis Questionnaire-Revised (CFQ-R) application calculates the score derived from the CFQ-R, on a 0-100 scale with higher scores indicating better HRQoL.
Change in Patient Health Questionnaire-9 (PHQ-9) Score | Baseline, 12 weeks
  The PHQ-9 measures severity of depression. Potential scores may range from 0 - 27 with higher scores indicating more severe depression.

SECONDARY OUTCOMES:
Change in nasal mucous biomarkers. | Baseline, 12 weeks
  A small strip of Leukosorb paper will be placed in the nostril to collect nasal mucous. The strips will be tested for the present of inflammatory markers including IL-4, IL-6, IL-8, TNF-alpha, IL-1B, Neutrophil elastase levels. The presence of inflammatory markers may indicate the return of neutrophilic infiltration.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Illing, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health, Indianapolis, Indiana, United States